CLINICAL TRIAL: NCT00133718
Title: Asker and Baerum Cardiovascular Diabetes Study
Brief Title: A 2 Year Trial of Patients With Type 2 Diabetes Focusing on Cardiovascular Diagnostics and Metabolic Control
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Asker & Baerum Hospital (Other)
Collaborators: Rikshospitalet University Hospital (Other); University Hospital, Aker (Other); Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Odd Erik Johansen, Study director, Asker & Baerum Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ABCD-study
Record Dates: First submitted 2005-08-23; First posted 2005-08-24 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 diabetes mellitus; Cardiovascular; Coronary artery disease; Glycemic control; Treatment; Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Coronary Artery Disease; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Patients were randomized to intensive care of standard care, outcomes were assessed by experts who where unaware of group allocation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Structured multi intervention (Other): Structured multi intervention to reach predefined glycemic and blood pressure goals as well as activity and weight goal
  Interventions: Drug: Combined lifestyle intervention and optimisation of pharmacological treatment
- Standard of care (Other): Standard care with or without structured care according to national guidelines
  Interventions: Drug: Combined lifestyle intervention and optimisation of pharmacological treatment

INTERVENTIONS:
Drug: Combined lifestyle intervention and optimisation of pharmacological treatment — 1. 6 months non-pharmacological treatment, 18 months with polypharmacy for glucose control (metformin, repaglinide/glimepiride, pioglitazone or insulin)
  2. standard care
  Other Names: Combination of drugs (predefined) to reach treatment targets

SUMMARY:
The purposes of this study are:

* to investigate the extent of cardiovascular complications in a representative cohort (n=135) of adult patients with type 2 diabetes;
* to examine if modern non-invasive assessment can replace invasive assessment;
* to determine the effects of a 6 month lifestyle interventional program on weight, glycemic control and lipids in 60 patients;
* to determine the effect of a 2-year prospective, randomised multi-interventional program (n=120) on cardiovascular risk, anthropometric measures and glycometabolic control; and
* to investigate inflammatory markers in this setting.

DETAILED DESCRIPTION:
As cardiovascular disease often is silent in type 2 diabetic patients, ways of detecting this early is of potential benefit, as is probably an aggressive treatment regimen trying to achieve goals for factors such as blood pressure, glycemic control, lipids, smoking, physical activity and weight.

This study compares traditional non-invasive tests such as stress-ecg, modern non-invasive tests such as holter-analysis, modern ECG analysis, stress-ecco cardiography and tissue Doppler against the gold standard today for assessing coronary artery disease, coronary angiography, in patients with type 2 diabetes and at least one cv-risk factor (i.e smoking, premature familial coronary artery disease (CAD)), hypertension) irrespective of symptoms or signs of CAD.

The participants are included in a randomized-control trial for 2 years where one arm receives standard treatment and one receives treatment after a multi-interventional program.

End-points include: glycemic control, lipid control, weight control, blood pressure control, and effects on inflammatory parameters.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Ages 18-75 years
* Men and women
* At least one cardiovascular risk factor (i.e hypertension, dyslipidemia, smoking/formerly smoker, premature familial coronary artery disease [CAD], microalbuminuria)
* Written informed consent given

Exclusion Criteria:

* Unwillingness
* Age < 18 or > 75 years
* Unstable cardiovascular condition
* Unstable medical condition

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2002-01; Primary Completion 2006-04 (Actual); Study Completion 2012-05-29 (Actual)

PRIMARY OUTCOMES:
Reduction in 10-year absolute CHD risk | 2-year

SECONDARY OUTCOMES:
Effects on cardiovascular events | 5-year
Effects on hospitalisations | 5-year
Effects on CV risk markers (HbA1c, lipids, blood pressure, inflammation, etc) | 2 years and 5 years
Effects on health related quality of life | 2 years and 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Odd E Johansen, MD, Principal Investigator — Asker and Baerum Hospital
Locations (1):
- Asker and Baerum Hospital, Medical Department, Rud, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ofstad AP, Johansen OE, Gullestad L, Birkeland KI, Orvik E, Fagerland MW, Urheim S, Aakhus S. Neutral impact on systolic and diastolic cardiac function of 2 years of intensified multi-intervention in type 2 diabetes: the randomized controlled Asker and Baerum Cardiovascular Diabetes (ABCD) study. Am Heart J. 2014 Sep;168(3):280-288.e2. doi: 10.1016/j.ahj.2014.03.026. Epub 2014 Jun 9. PMID 25173538
- [Background] Ulimoen GR, Ofstad AP, Endresen K, Gullestad L, Johansen OE, Borthne A. Low-dose CT coronary angiography for assessment of coronary artery disease in patients with type 2 diabetes--a cross-sectional study. BMC Cardiovasc Disord. 2015 Nov 14;15:147. doi: 10.1186/s12872-015-0143-9. PMID 26573616
- [Background] Johansen OE, Bjuro T, Endresen K, Blaasaas KG, Birkeland K, Aakhus S, Gullestad L. Heart rate adjustments and analysis of recovery patterns of ST-segment depression in type 2 diabetes. Int J Cardiol. 2008 Jun 23;127(1):129-32. doi: 10.1016/j.ijcard.2007.04.022. Epub 2007 May 25. PMID 17532067
- [Background] Johansen OE, Birkeland KI, Orvik E, Flesland O, Wergeland R, Ueland T, Smith C, Endresen K, Aukrust P, Gullestad L. Inflammation and coronary angiography in asymptomatic type 2 diabetic subjects. Scand J Clin Lab Invest. 2007;67(3):306-16. doi: 10.1080/00365510601045088. PMID 17454845
- [Background] Ofstad AP, Gullestad L, Orvik E, Aakhus S, Endresen K, Ueland T, Aukrust P, Fagerland MW, Birkeland KI, Johansen OE. Interleukin-6 and activin A are independently associated with cardiovascular events and mortality in type 2 diabetes: the prospective Asker and Baerum Cardiovascular Diabetes (ABCD) cohort study. Cardiovasc Diabetol. 2013 Aug 30;12:126. doi: 10.1186/1475-2840-12-126. PMID 23987834
- [Result] Johansen OE, Gullestad L, Blaasaas KG, Orvik E, Birkeland KI. Effects of structured hospital-based care compared with standard care for Type 2 diabetes-The Asker and Baerum Cardiovascular Diabetes Study, a randomized trial. Diabet Med. 2007 Sep;24(9):1019-27. doi: 10.1111/j.1464-5491.2007.02198.x. Epub 2007 May 17. PMID 17509068
- [Derived] Arora S, Ofstad AP, Ulimoen GR, Birkeland KI, Endresen K, Gullestad L, Johansen OE. Asymptomatic coronary artery disease in a Norwegian cohort with type 2 diabetes: a prospective angiographic study with intravascular ultrasound evaluation. Cardiovasc Diabetol. 2019 Mar 9;18(1):26. doi: 10.1186/s12933-019-0832-2. PMID 30851727
- [Derived] Ofstad AP, Ulimoen GR, Orvik E, Birkeland KI, Gullestad LL, Fagerland MW, Johansen OE. Long-term follow-up of a hospital-based, multi-intervention programme in type 2 diabetes mellitus: impact on cardiovascular events and death. J Int Med Res. 2017 Oct;45(5):1535-1552. doi: 10.1177/0300060517707674. Epub 2017 Jun 19. PMID 28627980